CLINICAL TRIAL: NCT00002167
Title: Photodynamic Therapy Clinical Trial For Cutaneous AIDS-Related Kaposi's Sarcoma Study Summary.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Solutions (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 261A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Skin Neoplasms; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Photochemotherapy; tin etiopurpurin; Radiation-Sensitizing Agents
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Skin Neoplasms; Acquired Immunodeficiency Syndrome | interventions — tin etiopurpurin

INTERVENTIONS:
Drug: Tin ethyl etiopurpurin

SUMMARY:
To determine the objective tumor response and remission rate of AIDS-related Kaposi's sarcomas (KS) following a single dose of tin ethyl etiopurpurin (SnET2) followed by photodynamic therapy (PDT). To determine the systemic and local toxicity, and morbidity safety profile of SnET2-PDT.

DETAILED DESCRIPTION:
All patients receive a single dose of SnET2 and are randomized to receive either PDT light treatment or no light treatment (control group). Patients are assessed prior to and at 4, 12 and 24 weeks following treatment, and are followed for 7 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documentation of at least one biopsy-confirmed KS lesion.
* A minimum of 4 and no more than 36 KS lesions.
* All eligible lesions must be bidimensionally measurable, treatable by surface (non-contact) light illumination, and <= 40 mm in diameter of the longest bidimensional axis.
* ACTG disease state T(0) L(0) or (1) S(0) or (1).
* Life expectancy greater than 6 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active opportunistic infection or condition except thrush or herpes simplex virus infections.
* Advanced KS tumor stages including the presence of tumor associated edema or ulceration, extensive oral KS, or KS in other non-nodal viscera.
* Hematopoietic dysfunction.
* Coagulation dysfunction.
* Hepatic dysfunction.
* Renal dysfunction.
* Cardiovascular dysfunction - Presence of significant coronary artery disease requiring current treatment or myocardial infarction.
* Pulmonary dysfunction.
* Sepsis.
* Known disorder of lipoprotein metabolism or clearance.

Patients with the following prior conditions are excluded:

* History of allergic or hypersensitivity reactions to light, egg proteins or egg yolks, history of porphyria, systemic lupus erythematosus or xeroderma pigmentosum.

Excluded within 7 days of therapy:

* Hematopoietic dysfunction.
* Coagulation dysfunction.
* Hepatic dysfunction.
* Renal dysfunction.

Excluded within 3 months of therapy:

* Pulmonary dysfunction.

Excluded within 6 months of therapy:

* Myocardial infarction.

Prior Medication:

Excluded:

* Intralesional chemotherapy within the past 12 weeks.
* Systemic chemotherapy or investigational drugs within the past 4 weeks.

Prior Treatment:

Excluded within 3 months prior to therapy:

* Local cryotherapy or surgery to study lesions.
* Systemic or topical photodynamic therapy agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Univ of Southern California / Los Angeles, Los Angeles, California
  - Cedars Sinai Med Ctr, Los Angeles, California
  - Univ of California / San Francisco / Dermatology, San Francisco, California
  - Health One - Rocky Mountain Cancer Ctr, Denver, Colorado
  - Buffalo Gen Hosp / PDT Ctr, Buffalo, New York
  - Thompson Cancer Survival Ctr, Knoxville, Tennessee